CLINICAL TRIAL: NCT00525785
Title: A Phase II Trial of Preoperative Chemotherapy and Chemoradiotherapy for Potentially Resectable Adenocarcinoma of the Stomach and Gastroesophageal Junction
Brief Title: Preoperative Chemo and Chemoradiotherapy for Adenocarcinoma of the Stomach and Gastroesophageal Junction (GEJ)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Sanofi-Synthelabo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0769; NCI-2010-00749 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-01

CONDITIONS: Stomach Cancer; Gastric Cancer
Keywords: Stomach Cancer; Gastric Cancer; Adenocarcinoma of the Stomach; Gastroesophageal Junction; Esophageal; Gastric; 5-Fluorouracil; 5-FU; Adrucil; Efudex; Folinic Acid; Oxaliplatin; Eloxatin; Chemoradiotherapy; Radiation; Radiotherapy; XRT
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 5-Fluorouracil + Folinic Acid + Oxaliplatin (Experimental): PreOp Chemotherapy: 2 cycles (each cycle consisting of 4 weeks or 2 treatments) of chemotherapy with oxaliplatin, folinic acid and infusional 5-FU (FOLFOX-48). Oxaliplatin 100 mg/m^2 over 2 hours on day 1, folinic acid intravenous (IV) at 200 mg/m^2 over 30 minutes on day 1, and 5-FU 2,200 mg/m^2 over 48 hours as continuous infusion by outpatient pump starting on day 1. This therapy, FOLFOX-48 repeated every 2 weeks x 4 (8 weeks of induction chemotherapy).
  PreOp Chemoradiotherapy begins 12 days after last dose of PreOp Chemo 5FU plus oxaliplatin; A total of 45 Gy (1.8 Gy fx/d) of radiotherapy concurrent to low-dose continuous infusion of 5-FU (300 mg/m^2/d Monday through Friday) & weekly oxaliplatin 45 mg/m^2 over 2 hours for 5 weeks (oxaliplatin administered on the first day of radiation week).
  Surgical resection 4-6 weeks after completion of chemoradiotherapy
  Interventions: Drug: 5-Fluorouracil; Drug: Folinic Acid; Drug: Oxaliplatin; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: 5-Fluorouracil — 2.2 Gm/m^2 By Vein Over 48 Hours On Days 1, 15, 29, and 43.
  Chemoradiotherapy: 300 mg/m2 a day Monday through Friday, by continuous infusion during radiation through an outpatient portable pump.
  Other Names: 5-FU; Adrucil; Efudex
Drug: Folinic Acid — 200 mg/m^2 by vein Over 30 Minutes On Days 1, 15, 29, and 43.
Drug: Oxaliplatin — 100 mg/m^2 By Vein Over 2 Hours On Days 1, 15, 29, and 43.
  Chemoradiotherapy: 45 mg/m^2 over 2 hours weekly for 5 weeks during radiation. (oxaliplatin should be administered on the first day of the radiation week).
  Other Names: Eloxatin
Radiation: Radiotherapy — 45 Gy (1.8 Gy fx/day) Monday through Friday, 12 days after the last dose of 5FU plus oxaliplatin and no later than 28 days.
  Other Names: XRT
Procedure: Surgery — 4-6 weeks after completion of chemoradiotherapy, restaged & surgical resection of the primary tumor and lymph nodes attempted.

SUMMARY:
The goal of this clinical research study is to learn if a combination of 5-FU, Folinic Acid and Oxaliplatin, given with radiation therapy, is effective in the treatment of gastric or gastroesophageal cancers that will be removed by surgery if possible. The safety of this combination therapy will also be studied.

DETAILED DESCRIPTION:
Oxaliplatin and 5-FU are chemotherapy drugs that are commonly used to treat certain kind of cancers. Folinic Acid (leucovorin) acts with 5-FU to increase cancer cell death.

Before treatment begins, you will be asked questions about your medical history and have a complete physical exam. You will have around 1 tablespoon of blood drawn for routine tests. You will have your height and weight measured. You will have a chest x-ray and an electrocardiogram (ECG - a test that measures the electrical activity of the heart). You will also have a chest x-ray, barium study of the upper gastrointestinal tract, and a CT scan to check the size and location of the tumor. Women who are able to have children must have a negative blood pregnancy test.

All patients will have had a routine upper gastrointestinal tract endoscopy and biopsy with endoscopic ultrasound examination prior to participating in this trial. However, once participating in this trial, the upper gastrointestinal tract endoscopy will be repeated prior to surgery. This procedure involves examination of the esophagus, stomach, and duodenum by a flexible tube. Biopsies will be taken as necessary.

You will receive treatment with 5-FU as an infusion into a vein using a continuous 24- hour portable pump. This will start on Day 1 and will continue for 48 hours. You will need to carry this pump with you at all times for 48 hours. The pump is about the size of a Sony Walkman®. You will also receive Oxaliplatin as an infusion into a vein over 2 hours on Day 1. Folinic Acid will be given as an infusion into a vein over 30 minutes on Day 1. You will have 12 days to recover between chemotherapy treatments. These drugs may be given to you as an outpatient. Treatment will be repeated on Day 15. Two 14-day treatment periods are called one cycle. You will receive up to 8 weeks of the above chemotherapy (2 cycles).

If the cancer gets worse or you experience intolerable side effects, you will be taken off the study and your doctor will discuss other treatment options with you.

Each week while you are receiving chemotherapy, around 1 tablespoon of blood will be drawn for routine tests.

Twelve days after you complete the second cycle of chemotherapy, you will begin to receive chemoradiotherapy (chemotherapy given at the same time as radiation therapy). Before chemoradiotherapy, you will be given a full physical, upper GI x-rays, about a tablespoon of blood will be drawn for routine blood tests, and if needed, a CT of the abdomen, chest and pelvis will be performed.

You will receive radiation therapy every weekday for a total of 25 sessions. During radiation therapy, 5-FU will be infused into your vein using a continuous infusion portable pump that you will carry with you day and night for up to 5 days (from Monday to Friday) of every week for 5 weeks. On Day 1 of radiation therapy each week, you will be given an infusion of Oxaliplatin into your vein over 2 hours for 5 weeks. During radiation therapy, you will be evaluated once a week and about one tablespoon of blood drawn for routine blood tests. Your doctor will discuss with you whether you will receive proton or x-ray radiation. If you receive proton radiation, it will be given in a building that is about a 5-minute drive from the M. D. Anderson radiation clinic.

If the cancer gets worse or you experience intolerable side effects, your treatment may be delayed or you may be taken off study and your doctor will discuss other treatment options with you.

Four to six weeks after the completion of chemoradiotherapy, the stage of the cancer will be evaluated. This includes drawing blood (about a tablespoon) for routine tests, chest x-ray, CT of the abdomen, chest, and pelvis (when necessary), upper GI endoscopy, and abdominal disease staging (if necessary).

When re-staging is complete, surgical removal of the primary tumor and lymph nodes will be attempted. All patients will be eligible for surgery. The J-tube will be left in your body for at least 8 weeks after the surgery to supplement your nutrition.

You will be asked to fill out side effect sheets throughout your participation in this research study. You will be asked questions regarding nausea, hair loss, fatigue, meals, and other questions regarding your daily activities.

Following this study, you will be asked to come for follow-up visits at M. D. Anderson at 3, 6, 9, and 12 months after surgery. You will then come in for visits every 6 months until Year 3, then once a year until Year 5. At these visits, you will have a full physical, about one tablespoon of blood drawn for routine tests, a chest x-ray, upper GI radiographs, upper GI endoscopy (every other visit) and CT of the abdomen (as needed).

This is an investigational study. Oxaliplatin is FDA approved and commercially available for the treatment of advanced colorectal cancer. Oxaliplatin is not approved in the US for the treatment of gastric cancer. 5-FU and folinic acid are commercially available drugs. The combination of these 3 drugs (Oxaliplatin + 5-FU + Folinic Acid) is investigational. A total of up to 58 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with potentially resectable adenocarcinoma of the stomach with histologic proof of adenocarcinoma, clinically staged T2-3, any N, M0 or T1N1M0 Gastric carcinoma may involve the gastroesophageal junction, however, the bulk of the tumor must be in the stomach (defined by radiographs, endoscopy, or endoscopic ultrasonography).
2. No prior major surgery of the stomach or radiation therapy to the stomach or immunotherapy or chemotherapy.
3. Patients must have a performance status of < 2 Zubrod scale.
4. Patients must have adequate bone marrow function (defined as peripheral absolute granulocyte count of >1,500/µL, and platelet count of > 100,000/µL), adequate liver function (bilirubin <= 1.5 mg/dl), and adequate renal function (creatinine <= 1.5 mg/dl).
5. Pretreatment evaluations must be done per the guidelines in Section 8.0.
6. A feeding jejunostomy must be inserted in all patients.
7. Patient must sign an informed consent prior to study entry.
8. Patient must be chronologic <= 75.

Exclusion Criteria:

1. Patients with T1N0 MO or T4 carcinoma documented by endoscopic ultrasonography.
2. Positive cytology of pleural, or pericardial effusion or patients with any peritoneal disease diagnosed by laparoscopy.
3. Biopsy proof of lymph node metastases outside the study field such as supraclavicular, mediastinal, or para-aortic nodes.
4. Evidence of metastatic disease to distant organs (biopsy is suggested for questionable findings).
5. Patients with cardiac disease graded as New York Heart Association Class III or IV, severe uncontrolled diabetes, hypertension, cerebrovascular disease, or infection.
6. Patients with diabetic neuropathy.
7. Abnormalities of mental status such that either the patient cannot fully comprehend the therapeutic implications of the protocol or comply with the requirements.
8. Presence of concurrent or previous malignancies in the past 5 years (except for resected squamous or basal cell carcinoma of the skin).
9. Pregnant women are excluded from study entry due to the potential teratogenic effects of the study treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2004-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: January 13, 2004 to October 25, 2010. All recruitment done at The University of Texas MD Anderson Cancer Center.
Period: Overall Study
Arm/Group | 5-Fluorouracil + Folinic Acid + Oxaliplatin
Started | 58
Completed | 55
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- 5-Fluorouracil + Folinic Acid + Oxaliplatin: FOLFOX-48 PreOp Chemotherapy (2 Cycles) with oxaliplatin, folinic acid & infusional 5-FU repeated every 2 weeks x 4 (8 weeks of induction chemotherapy). PreOp Chemoradiotherapy following PreOp Chemo 5FU plus oxaliplatin for total 45 Gy (1.8 Gy fx/d) of radiotherapy concurrent to low-dose continuous infusion of 5-FU (300 mg/m^2 for 5 days) & weekly oxaliplatin 45 mg/m^2 for 5 weeks (oxaliplatin administered on the first day of radiation week). Surgical resection 4-6 weeks after completion of chemoradiotherapy
Arm/Group | 5-Fluorouracil + Folinic Acid + Oxaliplatin
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 55.5 [29.0 to 74.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 45
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 58

OUTCOME MEASURES:

1. Primary Outcome: Complete Pathologic Response Rate
Description: The complete pathologic response (path CR) rate after treatment calculated as the percentage of participants with path CR out of the total participants, where the path CR is defined as absence of tumor cells in the surgical specimen and all registered participants are used in the denominator for calculating the path CR rate.
  Primary gastric carcinoma is not measurable by conventional criteria thus usual response criteria cannot be applied. The following criteria for response assessment applied: Pathologic Complete Response: Absence of tumor cells in the surgical specimen, 95% or more necrosis of the cancer; Complete Clinical Response: Absence of tumor on endoscopy, biopsy, cytology, or both.
Time Frame: Restaging and surgical resection at 4-6 weeks after completion of chemoradiotherapy, approximately at 16 weeks into treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 5-Fluorouracil + Folinic Acid + Oxaliplatin
Number analyzed (Participants) | 58
percentage of participants | 14 [6 to 25]

ADVERSE EVENTS:
Time Frame: Adverse event collection during 16 week+ treatment period using Common Toxicity Criteria (CTC) to score chemotherapy events and acute radiation (< 90 days) toxicities.
Description: Regular investigator assessment, regular laboratory testing, and routine questioning of participants during treatment and visits used for determination of adverse events.
Arm/Group | 5-Fluorouracil + Folinic Acid + Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 0/58
Serious Adverse Events (participants affected / at risk) | 4/58
Other Adverse Events (participants affected / at risk) | 42/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5-Fluorouracil + Folinic Acid + Oxaliplatin (N=58)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI-Stomach (Gastrointestinal disorders) | 4
Hyperbilrubinemia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Nausea Vomiting (Gastrointestinal disorders) | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
GI Bleed (Gastrointestinal disorders) | 4
Jejunostomy tube placement (planned procedure) (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 5-Fluorouracil + Folinic Acid + Oxaliplatin (N=58)
Anemia (Blood and lymphatic system disorders) | 26
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 14
Granulocytopenia (Blood and lymphatic system disorders) | 6
Increase ALT (Blood and lymphatic system disorders) | 6
Increase AST (Blood and lymphatic system disorders) | 7
Fatigue (General disorders) | 42
Myalgia (Musculoskeletal and connective tissue disorders) | 19
Neuropathy (Nervous system disorders) | 36
Nausea (Gastrointestinal disorders) | 40
Vomiting (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 31
Constipation (Gastrointestinal disorders) | 18
Dysphagaia (Gastrointestinal disorders) | 20
Reflux GERD (Gastrointestinal disorders) | 25
Anorexia (Gastrointestinal disorders) | 42
Stomatitis (Gastrointestinal disorders) | 17
Eyes red, Watery, Burning (Eye disorders) | 14
Skin Rash (Skin and subcutaneous tissue disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dizziness (Nervous system disorders) | 11
Insomnia (General disorders) | 29
Hand, Foot, Skin (Skin and subcutaneous tissue disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 8
J-tube pain (Gastrointestinal disorders) | 7
Substernal chest pain (Musculoskeletal and connective tissue disorders) | 3
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes